CLINICAL TRIAL: NCT06172348
Title: A PHASE 1, OPEN-LABEL STUDY IN HEALTHY PARTICIPANTS TO INVESTIGATE THE PHARMACOKINETICS OF RITLECITINIB FOLLOWING SINGLE ORAL ADMINISTRATION OF MODIFIED RELEASE FORMULATIONS UNDER FED AND FASTED CONDITIONS
Brief Title: A Study to Learn About Three Forms of The Study Medicine (Ritlecitinib) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7981086; 2023-505603-23-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Adults
MeSH Terms: interventions — PF-06651600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment Sequence 1 (Experimental): Ritlecitinib 100 mg solution (fasted, Period 1), followed by ritlecitinib 100 mg MR capsule 1 (fasted, Period 2), followed by ritlecitinib 100 mg MR capsule 2 (fasted, Period 3), and followed by ritlecitinib 100 mg MR capsule 1 (fed, Period 4)
  Interventions: Drug: Ritlecitinib
- Treatment Sequence 2 (Experimental): Ritlecitinib 100 mg MR capsule 1 (fasted, Period 1), followed by ritlecitinib 100 mg MR capsule 2 (fasted, Period 2), followed by ritlecitinib 100 mg solution (fasted, Period 3), and followed by ritlecitinib 100 mg MR capsule 1 (fed, Period 4)
  Interventions: Drug: Ritlecitinib
- Treatment Sequence 3 (Experimental): Ritlecitinib 100 mg MR capsule 2 (fasted, Period 1), followed by ritlecitinib 100 mg solution (fasted, Period 2), followed by ritlecitinib 100 mg MR capsule 1 (fasted, Period 3), and followed by ritlecitinib 100 mg MR capsule 1 (fed, Period 4)
  Interventions: Drug: Ritlecitinib
- Treatment Sequence 4 (Experimental): Ritlecitinib 100 mg solution (fasted, Period 1), followed by ritlecitinib 100 mg MR capsule 1 (fasted, Period 2), followed by ritlecitinib 100 mg MR capsule 2 (fasted, Period 3), and followed by ritlecitinib 100 mg MR capsule 2 (fed, Period 4)
  Interventions: Drug: Ritlecitinib
- Treatment Sequence 5 (Experimental): Ritlecitinib 100 mg MR capsule 1 (fasted, Period 1), followed by ritlecitinib 100 mg MR capsule 2 (fasted, Period 2), followed by ritlecitinib 100 mg solution (fasted, Period 3), and followed by ritlecitinib 100 mg MR capsule 2 (fed, Period 4)
  Interventions: Drug: Ritlecitinib
- Treatment Sequence 6 (Experimental): Ritlecitinib 100 mg MR capsule 2 (fasted, Period 1), followed by ritlecitinib 100 mg solution (fasted, Period 2), followed by ritlecitinib 100 mg MR capsule 1 (fasted, Period 3), and followed by ritlecitinib 100 mg MR capsule 2 (fed, Period 4)
  Interventions: Drug: Ritlecitinib

INTERVENTIONS:
Drug: Ritlecitinib — Ritlecitinib 100 milligrams (mg) will be provided as either solution or capsule formulation (2 capsules of 50 mg)
  Other Names: PF-06651600

SUMMARY:
The purpose of this study is to compare if three forms of study medicine (called ritlecitinib) get processed differently in healthy adults.

This study is seeking healthy participants who have:

* Aged 18 years or older;
* male or female who are healthy as determined by medical assessment;
* BMI of 16-32 kg/m2, and a total body weight >45 kg (99 lb).

All participants in this study will receive a ritlecitinib oral dose in three different forms (solution, capsule 1 and capsule 2).

The study will take up to 2.5 months, including the screening period and follow-up phone call. Participants will have to stay at the study clinic for at least 13 days. There will be 4 periods in total for this study. On day 1 of each period, participants will take one form of Riltecitinib without food for the first three periods and with food for the last period. Participants will have blood samples taken both before and after taking ritlecitinib. A follow-up phone call will be made at 28 to 35 days after the last study period.

DETAILED DESCRIPTION:
Ritlecitinib is a covalent and irreversible inhibitor of JAK3 with high selectivity over the other JAK isoforms (JAK1, JAK2, and TYK2). Ritlecitinib also inhibits irreversibly the TEC family kinases with selectivity over the broader human kinome. Treatment with ritlecitinib is expected to inhibit the inflammatory pathways mediated by IL 7, IL 15 and IL 21, all implicated in UC, CD, AA, RA, and vitiligo and therefore under development in these indications. Moreover, due to lack of activity against the other JAK isoforms, ritlecitinib is expected to spare immunoregulatory cytokines such as IL 10, IL 27 and IL 35, which are critical to the maintenance of immunosuppressive functions and immune homeostasis.

This study aims to investigate the pharmacokinetics (PK) and relative bioavailability of 2 new modified release (MR) capsule formulations of ritlecitinib, MR1 (release duration: 6-8 hours) and MR2 (release duration:13 15 hours) as single doses in fasted and fed conditions.

This is a single dose, open-label, randomized, 4-period, 6-sequence crossover study in a single cohort of approximately 12 healthy participants randomized to one of the sequences (containing 1 solution and 2 modified release [MR1 and MR2] capsule formulations of ritlecitinib) described in the table below. The first 3 periods are under fasted condition and the fourth period is under fed condition to investigate the effect of food on the PK of MR1 and MR2.

For a given participant, the total study duration from screening to follow-up phone call will be between approximately 8 to 11 weeks.

Screening will occur within 28 days prior to the first dose of the study intervention. Each participant will go through Periods 1 through 4 and dosing in each treatment period will be separated by at least 3 days to minimize any carryover effect.

Venous PK blood samples for PK analysis will be collected pre-dose and post-dose in each period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
2. BMI of 16-32 kg/m2, and a total body weight >45 kg (99 lb).
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Capable of giving signed informed consent

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Participants with the acute or chronic infections or infection history
3. History of febrile illness within 5 days prior to the first dose of study intervention.
4. History of any lymphoproliferative disorder such as EBV related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs or symptoms suggestive of current lymphatic or lymphoid disease.
5. Known present or a history of malignancy other than a successfully treated or excised nonmetastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
6. History of active or latent Mycobacterium TBA: participant who is currently being treated for active or latent Mycobacterium TB infection or has a history of Mycobacterium TB must be excluded from the study.
7. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981086

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received treatment in Period 1, 2 or 3 under fasted condition and in Period 4 under fed condition.
Groups:
- Treatment Sequence 1: A Then B Then C Then B (Fed): Participants were randomized to receive ritlecitinib 100 milligrams (mg) single oral dose as oral solution [A] in fasted state on Day 1 of Period 1; then ritlecitinib 100 mg (2*50 mg) single oral dose as modified release1 (MR1) capsules [B] in fasted state on Day 1 of Period 2; then ritlecitinib 100 mg (2*50 mg) single oral dose as MR2 capsules [C] in fasted state on Day 1 of Period 3; and then ritlecitinib 100 mg (2*50 mg) single oral dose as MR1 capsules [B] in fed state of Period 4. Between 2 doses of consecutive periods there was a gap of at least 48 hours.
- Treatment Sequence 2: B Then C Then A Then B (Fed): Participants were randomized to receive ritlecitinib 100 mg (2*50 mg) single oral dose as MR1 capsules [B] in fasted state on Day 1 of Period 2; then ritlecitinib 100 mg (2*50 mg) single oral dose as MR2 capsules [C] in fasted state on Day 1 of Period 3; then ritlecitinib 100 mg single oral dose as oral solution [A] in fasted state on Day 1 of Period 1; and then ritlecitinib 100 mg (2*50 mg) single oral dose as MR1 capsules [B] in fed state of Period 4. Between 2 doses of consecutive periods there was a gap of at least 48 hours.
- Treatment Sequence 3: C Then A Then B Then B (Fed): Participants were randomized to receive ritlecitinib 100 mg (2*50 mg) single oral dose as MR2 capsules [C] in fasted state on Day 1 of Period 3; then ritlecitinib 100 mg single oral dose as oral solution [A] in fasted state on Day 1 of Period 1; then ritlecitinib 100 mg (2*50 mg) single oral dose as MR1 capsules [B] in fasted state on Day 1 of Period 2; and then ritlecitinib 100 mg (2*50 mg) single oral dose as MR1 capsules [B] in fed state of Period 4. Between 2 doses of consecutive periods there was a gap of at least 48 hours.
- Treatment Sequence 4: A Then B Then C Then C (Fed): Participants were randomized to receive ritlecitinib 100 mg single oral dose as oral solution [A] in fasted state on Day 1 of Period 1; then ritlecitinib 100 mg (2*50 mg) single oral dose as MR1 capsules [B] in fasted state on Day 1 of Period 2; then ritlecitinib 100 mg (2*50 mg) single oral dose as MR2 capsules [C] in fasted state on Day 1 of Period 3; and then ritlecitinib 100 mg (2*50 mg) single oral dose as MR2 capsules [C] in fed state of Period 4. Between 2 doses of consecutive periods there was a gap of at least 48 hours.
- Treatment Sequence 5: B Then C Then A Then C (Fed): Participants were randomized to receive ritlecitinib 100 mg (2*50 mg) single oral dose as MR1 capsules [B] in fasted state on Day 1 of Period 2; then ritlecitinib 100 mg (2*50 mg) single oral dose as MR2 capsules [C] in fasted state on Day 1 of Period 3; then ritlecitinib 100 mg single oral dose as oral solution [A] in fasted state on Day 1 of Period 1; and then ritlecitinib 100 mg (2*50 mg) single oral dose as MR2 capsules [C] in fed state of Period 4. Between 2 doses of consecutive periods there was a gap of at least 48 hours.
- Treatment Sequence 6: C Then A Then B Then C (Fed): Participants were randomized to receive ritlecitinib 100 mg (2*50 mg) single oral dose as MR2 capsules [C] in fasted state on Day 1 of Period 3; then ritlecitinib 100 mg single oral dose as oral solution [A] in fasted state on Day 1 of Period 1; then ritlecitinib 100 mg (2*50 mg) single oral dose as MR1 capsules [B] in fasted state on Day 1 of Period 2; and then ritlecitinib 100 mg (2*50 mg) single oral dose as MR2 capsules [C] in fed state of Period 4. Between 2 doses of consecutive periods there was a gap of at least 48 hours.
Period: Treatment Period 1
Arm/Group | Treatment Sequence 1: A Then B Then C Then B (Fed) | Treatment Sequence 2: B Then C Then A Then B (Fed) | Treatment Sequence 3: C Then A Then B Then B (Fed) | Treatment Sequence 4: A Then B Then C Then C (Fed) | Treatment Sequence 5: B Then C Then A Then C (Fed) | Treatment Sequence 6: C Then A Then B Then C (Fed)
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Treatment Sequence 1: A Then B Then C Then B (Fed) | Treatment Sequence 2: B Then C Then A Then B (Fed) | Treatment Sequence 3: C Then A Then B Then B (Fed) | Treatment Sequence 4: A Then B Then C Then C (Fed) | Treatment Sequence 5: B Then C Then A Then C (Fed) | Treatment Sequence 6: C Then A Then B Then C (Fed)
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 1 | 2 | 2 | 2
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Treatment Sequence 1: A Then B Then C Then B (Fed) | Treatment Sequence 2: B Then C Then A Then B (Fed) | Treatment Sequence 3: C Then A Then B Then B (Fed) | Treatment Sequence 4: A Then B Then C Then C (Fed) | Treatment Sequence 5: B Then C Then A Then C (Fed) | Treatment Sequence 6: C Then A Then B Then C (Fed)
Started | 2 | 2 | 1 | 2 | 2 | 2
Completed | 2 | 2 | 1 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Treatment Sequence 1: A Then B Then C Then B (Fed) | Treatment Sequence 2: B Then C Then A Then B (Fed) | Treatment Sequence 3: C Then A Then B Then B (Fed) | Treatment Sequence 4: A Then B Then C Then C (Fed) | Treatment Sequence 5: B Then C Then A Then C (Fed) | Treatment Sequence 6: C Then A Then B Then C (Fed)
Started | 2 | 2 | 1 | 2 | 2 | 2
Completed | 2 | 2 | 1 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Sequence 1: A Then B Then C Then B (Fed): Participants were randomized to receive ritlecitinib 100 mg single oral dose as oral solution [A] in fasted state on Day 1 of Period 1; then ritlecitinib 100 mg (2*50 mg) single oral dose as MR1 capsules [B] in fasted state on Day 1 of Period 2; then ritlecitinib 100 mg (2*50 mg) single oral dose as MR2 capsules [C] in fasted state on Day 1 of Period 3; and then ritlecitinib 100 mg (2*50 mg) single oral dose as MR1 capsules [B] in fed state of Period 4. Between 2 doses of consecutive periods there was a gap of at least 48 hours.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1: A Then B Then C Then B (Fed) | Treatment Sequence 2: B Then C Then A Then B (Fed) | Treatment Sequence 3: C Then A Then B Then B (Fed) | Treatment Sequence 4: A Then B Then C Then C (Fed) | Treatment Sequence 5: B Then C Then A Then C (Fed) | Treatment Sequence 6: C Then A Then B Then C (Fed) | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 2 | 1 | 2 | 10
  >=65 years | 0 | 0 | 1 | 0 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Male | 2 | 2 | 2 | 1 | 2 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 2 | 1 | 2 | 2 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 1 | 1 | 4
  White | 2 | 2 | 1 | 1 | 1 | 1 | 8
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Ritlecitinib: MR Capsules vs Oral Solution Under Fasted Condition
Time Frame: For oral solution: Pre-dose (0 hours), 0.5, 1, 2, 3, 4, 6, 10, 12 and 24 hours post-dose on Day 1 of Period 1, 2 or 3; for MR1 and MR2 capsules: Pre-dose (0 hours), 1, 2, 3, 4, 6, 10, 12,16, 24, 36 and 48 hours post-dose on Day 1 of Period 1, 2 or 3
Population: Pharmacokinetic (PK) parameter set included all participants who had at least 1 PK parameter of interest quantified in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Groups:
- Ritlecitinib 100 mg Oral Solution (Fasted): Participants received Ritlecitinib 100 mg as oral solution under fasted conditions on Day 1 of either Period 1, 2, or 3.
- Ritlecitinib 100 mg MR1 Capsule (Fasted): Participants received Ritlecitinib 100 mg as oral MR1 capsules under fasted conditions on Day 1 of either Period 1, 2, or 3.
- Ritlecitinib 100 mg MR2 Capsule (Fasted): Participants received Ritlecitinib 100 mg as oral MR2 capsules under fasted conditions on Day 1 of either Period 1, 2, or 3.
Arm/Group | Ritlecitinib 100 mg Oral Solution (Fasted) | Ritlecitinib 100 mg MR1 Capsule (Fasted) | Ritlecitinib 100 mg MR2 Capsule (Fasted)
Number analyzed (Participants) | 12 | 11 | 12
Nanogram per milliliter (ng/mL) | 671.6 (24) | 145.1 (25) | 84.96 (25)
Statistical Analysis 1: Comparison: Ritlecitinib 100 mg Oral Solution (Fasted) vs Ritlecitinib 100 mg MR1 Capsule (Fasted); A mixed effect model was used with sequence, period and treatment as fixed effects and participant with sequence as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 21.89, 90% CI 2-sided [19.31 to 24.80] — Ratios (Test/Reference) and 90 percent (%) confidence intervals were expressed as percentages. Test = MR1 capsule; Reference = Oral solution
Statistical Analysis 2: Comparison: Ritlecitinib 100 mg Oral Solution (Fasted) vs Ritlecitinib 100 mg MR2 Capsule (Fasted); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 12.65, 90% CI 2-sided [11.21 to 14.27] — Ratios (Test/Reference) and 90% confidence intervals were expressed as percentages. Test = MR2 capsule; Reference = Oral solution

2. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero (0) Extrapolated to Infinite Time (AUCinf) of Ritlecitinib: MR Capsules vs Oral Solution Under Fasted Condition
Description: AUCinf was calculated as AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 1
Population: PK parameter set included all participants who had at least 1 PK parameter of interest quantified in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*Hour per milliliter (ng*hr/mL)
Arm/Group | Ritlecitinib 100 mg Oral Solution (Fasted) | Ritlecitinib 100 mg MR1 Capsule (Fasted) | Ritlecitinib 100 mg MR2 Capsule (Fasted)
Number analyzed (Participants) | 12 | 11 | 12
Nanogram*Hour per milliliter (ng*hr/mL) | 1261 (23) | 1067 (28) | 970.6 (22)
Statistical Analysis 1: Comparison: Ritlecitinib 100 mg Oral Solution (Fasted) vs Ritlecitinib 100 mg MR1 Capsule (Fasted); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 86.49, 90% CI 2-sided [79.11 to 94.54] — Ratios (Test/Reference) and 90% confidence intervals were expressed as percentages. Test = MR1 capsule; Reference = Oral solution
Statistical Analysis 2: Comparison: Ritlecitinib 100 mg Oral Solution (Fasted) vs Ritlecitinib 100 mg MR2 Capsule (Fasted); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 76.99, 90% CI 2-sided [70.65 to 83.90] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Cmax of Ritlecitinib: MR Capsules Under Fed vs Fasted Condition
Time Frame: Pre-dose (0 hours), 1, 2, 3, 4, 6, 10, 12,16, 24, 36 and 48 hours post-dose on Day 1 of Period 1, 2, 3 (for fasted) or 4 (for fed)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Groups:
- Ritlecitinib 100 mg MR1 Capsule (Fed): Participants received Ritlecitinib 100 mg as oral MR1 capsules under fed conditions on Day 1 of Period 4.
- Ritlecitinib 100 mg MR2 Capsule (Fed): Participants received Ritlecitinib 100 mg as oral MR2 capsules under fed conditions on Day 1 of Period 4.
Arm/Group | Ritlecitinib 100 mg MR1 Capsule (Fasted) | Ritlecitinib 100 mg MR2 Capsule (Fasted) | Ritlecitinib 100 mg MR1 Capsule (Fed) | Ritlecitinib 100 mg MR2 Capsule (Fed)
Number analyzed (Participants) | 11 | 12 | 5 | 6
Nanogram per milliliter (ng/mL) | 145.1 (25) | 84.96 (25) | 177.1 (16) | 112.0 (14)
Statistical Analysis 1: Comparison: Ritlecitinib 100 mg MR1 Capsule (Fasted) vs Ritlecitinib 100 mg MR1 Capsule (Fed); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 123.92, 90% CI 2-sided [105.16 to 146.02] — Ratios (Test/Reference) and 90% confidence intervals were expressed as percentages. Test = MR1 capsule (fed); Reference = MR1 capsule (fasted)
Statistical Analysis 2: Comparison: Ritlecitinib 100 mg MR2 Capsule (Fasted) vs Ritlecitinib 100 mg MR2 Capsule (Fed); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 129.79, 90% CI 2-sided [111.51 to 151.06] — Ratios (Test/Reference) and 90% confidence intervals were expressed as percentages. Test = MR2 capsule (fed); Reference = MR2 capsule (fasted)

4. Secondary Outcome: AUCinf of Ritlecitinib: MR Capsules Under Fed vs Fasted Condition
Description: as for outcome 2
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*Hour per milliliter (ng*hr/ mL)
Arm/Group | Ritlecitinib 100 mg MR1 Capsule (Fasted) | Ritlecitinib 100 mg MR2 Capsule (Fasted) | Ritlecitinib 100 mg MR1 Capsule (Fed) | Ritlecitinib 100 mg MR2 Capsule (Fed)
Number analyzed (Participants) | 11 | 12 | 5 | 6
Nanogram*Hour per milliliter (ng*hr/ mL) | 1067 (28) | 970.6 (22) | 1168 (20) | 1036 (15)
Statistical Analysis 1: Comparison: Ritlecitinib 100 mg MR1 Capsule (Fasted) vs Ritlecitinib 100 mg MR1 Capsule (Fed); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 107.48, 90% CI 2-sided [96.46 to 119.76] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Ritlecitinib 100 mg MR2 Capsule (Fasted) vs Ritlecitinib 100 mg MR2 Capsule (Fed); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 109.63, 90% CI 2-sided [99.19 to 121.17] — [estimate comment as in outcome 3, analysis 2]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: From start of study treatment up to 35 days after administration of last dose of study intervention (maximum up to 45 days)
Population: Safety analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 100 mg Oral Solution (Fasted) | Ritlecitinib 100 mg MR1 Capsule (Fasted) | Ritlecitinib 100 mg MR2 Capsule (Fasted) | Ritlecitinib 100 mg MR1 Capsule (Fed) | Ritlecitinib 100 mg MR2 Capsule (Fed)
Number analyzed (Participants) | 12 | 11 | 12 | 5 | 6
Participants | 3 | 5 | 3 | 0 | 1

6. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormalities
Description: Laboratory parameters included: Hematology: lymphocytes/leukocytes, eosinophils/leukocytes greater than (>) 1.2*upper limit of normal (ULN) (percent [%]), neutrophils/leukocytes less than (<) 0.8*lower limit of normal (LLN) (%); Urinalysis: urine hemoglobin, nitrite greater than or equal to (>=) 1, bacteria > 20 (per high power field [/HPF]). Clinical significance was judged by investigator.
Time Frame: From start of study treatment up to Day 3 of Period 4 (maximum up to Day 12, each Period = 3 days)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Groups:
- Ritlecitinib 100 mg (MR2 Capsule) Fed: Participants received Ritlecitinib 100 mg as oral MR2 capsules under fed conditions on Day 1 of Period 4.
Arm/Group | Ritlecitinib 100 mg Oral Solution (Fasted) | Ritlecitinib 100 mg MR1 Capsule (Fasted) | Ritlecitinib 100 mg MR2 Capsule (Fasted) | Ritlecitinib 100 mg MR1 Capsule (Fed) | Ritlecitinib 100 mg (MR2 Capsule) Fed
Number analyzed (Participants) | 12 | 11 | 12 | 5 | 6
Participants | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate (PR) were measured in a supine position. Criteria for vital signs included: SBP: value less than (<) 90 millimeter of mercury (mmHg), change greater than or equal to (>=) 30 mmHg decrease, change >= 30 mmHg increase; DBP: value < 50 mmHg, change >= 20 mmHg decrease, change >= 20 mmHg increase; PR: value < 40 beats per minute (bpm), value > 120 bpm. Clinical significance was judged by investigator.
Time Frame: From start of study treatment up to Day 3 of Period 4 (maximum up to Day 12, each Period = 3 days)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 100 mg Oral Solution (Fasted) | Ritlecitinib 100 mg MR1 Capsule (Fasted) | Ritlecitinib 100 mg MR2 Capsule (Fasted) | Ritlecitinib 100 mg MR1 Capsule (Fed) | Ritlecitinib 100 mg (MR2 Capsule) Fed
Number analyzed (Participants) | 12 | 11 | 12 | 5 | 6
Participants | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Standard 12 lead ECGs were obtained with the participant in a supine position after at least 5 minutes of rest using an ECG machine that automatically calculated the heart rate and measured PR interval, QT, corrected QT (Fridericia method) (QTcF) and QRS intervals. Clinical significance was judged by investigator.
Time Frame: From start of study treatment up to Day 3 of Period 4 (maximum up to Day 12, each Period = 3 days)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 100 mg Oral Solution (Fasted) | Ritlecitinib 100 mg MR1 Capsule (Fasted) | Ritlecitinib 100 mg MR2 Capsule (Fasted) | Ritlecitinib 100 mg MR1 Capsule (Fed) | Ritlecitinib 100 mg MR2 Capsule (Fed)
Number analyzed (Participants) | 12 | 11 | 12 | 5 | 6
Participants | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 35 days after administration of last dose of study intervention (maximum up to 45 days)
Description: Safety analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Groups:
- Ritlecitinib 100 mg MR1 Capsules (Fasted): Participants received Ritlecitinib 100 mg as oral MR1 capsules under fasted conditions on Day 1 of either Period 1, 2, or 3.
- Ritlecitinib 100 mg MR2 Capsules (Fasted): Participants received Ritlecitinib 100 mg as oral MR2 capsules under fasted conditions on Day 1 of either Period 1, 2, or 3.
- Ritlecitinib 100 mg MR1 Capsules (Fed): Participants received Ritlecitinib 100 mg as oral MR1 capsules under fed conditions on Day 1 of Period 4.
- Ritlecitinib 100 mg MR2 Capsules (Fed): Participants received Ritlecitinib 100 mg as oral MR2 capsules under fed conditions on Day 1 of Period 4.
Arm/Group | Ritlecitinib 100 mg Oral Solution (Fasted) | Ritlecitinib 100 mg MR1 Capsules (Fasted) | Ritlecitinib 100 mg MR2 Capsules (Fasted) | Ritlecitinib 100 mg MR1 Capsules (Fed) | Ritlecitinib 100 mg MR2 Capsules (Fed)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/12 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/12 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 3/12 | 5/11 | 3/12 | 0/5 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ritlecitinib 100 mg Oral Solution (Fasted) (N=12) | Ritlecitinib 100 mg MR1 Capsules (Fasted) (N=11) | Ritlecitinib 100 mg MR2 Capsules (Fasted) (N=12) | Ritlecitinib 100 mg MR1 Capsules (Fed) (N=5) | Ritlecitinib 100 mg MR2 Capsules (Fed) (N=6)
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT06172348/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT06172348/SAP_001.pdf